CLINICAL TRIAL: NCT04276194
Title: Feasibility of Vertebral Body Sparing Intensity Modulated Proton Therapy Craniospinal Irradiation With in Vivo Range Verification in Growing Children
Brief Title: Vertebral Body Sparing Craniospinal Irradiation for Pediatric Patients With Cancer of the Central Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Bree Eaton, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00113121; NCI-2019-05118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA138292 (NIH); RAD4737-19 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2020-01-27; First posted 2020-02-19 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Malignant Central Nervous System Neoplasm
Keywords: Craniospinal; Proton Therapy; Pediatric
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (intensity modulated proton therapy) (Experimental): Patients undergo intensity modulated proton therapy once daily over 30 fractions and also undergo MRI over 20 minutes during fractions 7, 13, 20, and 30 of radiation in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Intensity-Modulated Proton Therapy; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Intensity-Modulated Proton Therapy — Undergo intensity modulated proton therapy
  Other Names: IMPT
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This trial studies the feasibility of using intensity modulated proton therapy to deliver craniospinal irradiation while avoiding the bones of the vertebral column. Intensity modulated proton therapy is an advanced radiation therapy modality that uses high energy protons to kill cancer cells and shrink tumors, and may reduce the side effects of treatment by reducing radiation exposure to the spinal column.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the feasibility and safety of using intensity modulated proton therapy to deliver vertebral body sparing craniospinal irradiation in growing children.

Ia. To report the dose received to the vertebral bodies and the dose gradient/heterogeneity within the vertebral body.

Ib. To document, using weekly cone beam computed tomography (CT) of the cervical and lumbar spine, delivered dose in comparison with planned dose after accounting for any errors in patient positioning.

II. To evaluate acute toxicity of vertebral body sparing (VBS) craniospinal irradiation (CSI).

IIa. To report absolute lymphocyte counts over time and occurrence of grade 3-4 hematological toxicity.

IIb. To report the incidence and severity of any grade esophagitis during or within 4 weeks of radiation therapy.

III. To evaluate the feasibility of magnetic resonance imaging (MRI) imaging during CSI therapy as in vivo proton range verification.

IIIa. To demonstrate the feasibility of completing interim non-contrast MRIs of the spine during treatment.

IIIb. To characterize the earliest time point at which radiation induced bone marrow changes can be detected in children receiving proton CSI.

OUTLINE:

Patients undergo intensity modulated proton therapy once daily over 30 fractions and also undergo MRI over 20 minutes during fractions 7, 13, 20, and 30 of radiation in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients are followed up at 4 weeks and then every 3-12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of central nervous system malignancy requiring craniospinal irradiation.
* Signed informed consent and assent when indicated.

Exclusion Criteria:

* Any contraindication to undergoing MRI (ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial cardiac valves or devices, electrical implants such as cardiac pacemakers or perfusion pumps). Metal fragments, shrapnel, or tattoos near the eye.
* Any major uncontrolled or poorly controlled current illness that would limit compliance with study requirements.
* Pregnant females are excluded. Females of childbearing age/menstruating must confirm that either they are not sexually active or have a negative pregnancy test prior to initiation of radiation therapy.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of acute hematologic toxicity | Up to 2 years
  Will be graded according to Common Terminology Criteria for Adverse Events version 5.0.
Dose delivered to vertebral bodies and quality assurance of treatment plans | Up to 2 years
  Multiple measurements will be aggregated to arrive at one reported value when toxicities are graded (1-5). Dose statistics are in units of Gy or may be %
Bone marrow changes on MRI | At baseline, and fractions 7, 13, 20, and 30 of radiation therapy
  Will be quantitatively and qualitatively analyzed in relationship to the proton dose distribution

CONTACTS AND LOCATIONS:
Overall Officials: Bree R Eaton, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia

DOCUMENTS (1):
  • Informed Consent Form (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT04276194/ICF_000.pdf